CLINICAL TRIAL: NCT05482490
Title: A Novel Hygienic Maintenance Protocol for Implant Supported Hybrid Prosthesis. Prospective Clinical and Microbiological Outcomes
Brief Title: Maintenance Protocol for Implant Supported Hybrid Prosthesis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Assistant Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Perio4
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Implant Infection
Keywords: Dental Implants; Hybrid prosthesis; Supportive therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IFCDPprotocol (Experimental): Patients subjected to the novel implant-supported fixed complete dental prostheses maintenance protocol
  Interventions: Procedure: Maintenance protocol for the hygiene of implant supported prosthesis

INTERVENTIONS:
Procedure: Maintenance protocol for the hygiene of implant supported prosthesis — Sequence of phases that include the hygiene and cleaning of the prosthesis and the implants, the motivation of the patients and reinforcement of oral hygiene.

SUMMARY:
The study we intend to carry out aims to analyze the clinical and microbiological effects of a new maintenance protocol for implant-supported hybrid prostheses.

The maintenance protocol we propose is based on a sequence of phases that include not only the hygiene and cleaning of the prosthesis and the implants, but also the motivation and reinforcement of oral hygiene through iconographic aid (intraoral photographs of the patient).

The proposed hygiene protocol is based on a meticulous preliminary plaque disclosure, followed by a full mouth decontamination of all intraoral mucosae, a decontamination of the secondary components, specific intrasulcular decontamination of the implants depending on whether there are probes greater than or less than 5mm and finally, a decontamination and hygiene of the hybrid prosthesis, all with the help of erythritol powders and the different settings of the AirFlow Prophylaxis Master EMS (Electro Medical Systems S.A., Nyon, Switzerland) device.

Clinical parameters such as plaque index (PlI), probing depth (PD), bleeding on probing (BOP) and peri-implant suppuration (PS) will be recorded immediately after removal of the prosthesis and at one month of follow-up.

The collection of the microbiological sample will be carried out according to the following procedures: the implant will be isolated by suction and the use of cotton rolls, in order to avoid contamination of saliva. Four sterile endodontic paper points will be inserted into the peri-implant sulcus of each implant, placing them in the mesial, distal, lingual/palatal and buccal sites and removed after 30 seconds with tweezers by placing them in a sterile plastic tube which will be sealed immediately. The same procedure will be performed for each implant.

Once the operation is completed, the tubes of each patient (one for each implant and each containing 4 paper points) will be sent for microbiological analysis. The samples will be sent to the Microbiology Laboratory of the Department of Surgical Sciences of the University of Cagliari, in order to analyze the presence of bacteria ofn the peri-implant sulci. DNA from crevicular fluid samples will then be isolated by centrifugation and analyzed by PCR (polymerase chain reaction). This biomolecular technique is based on an enzymatic reaction, in which a heat-resistant DNA polymerase (Taq Polymerase) catalyzes the specific amplification of known DNA sequences. This procedure will be performed before the hygiene protocol, immediately after and at one month of follow-up.

Power analysis was employed to determine the sample size by using a .05 significance level and a power of 90% based on an effect size of 0.25. Sample size of a minimum of 130 implants (approximately 25/30 patients carrying implant supported hybrid prostheses) is required to detect significant difference between the parameters measured at the different time points using repeated measures ANOVA, however the recruitment of patients will continue through the entire first period of the execution program with no limitations even after reaching the predetermined number

DETAILED DESCRIPTION:
The study population will consist of patients presenting at the periodontology departments of the Universities of Cagliari and who need maintenance for implant-supported hybrid prostheses.

Patients will be excluded from the study if affected by chronic bronchitis or asthma and major systemic illnesses (i.e. diabetes mellitus, cancer, HIV, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy). Intake of antibiotics or other medication taken within the previous 28 days that may affect the outcome of the study will prevent inclusion in the study as well as confirmed or suspected intolerance to erythritol or chlorhexidine.

The implant-supported fixed complete dental prostheses maintenance protocol will consist in the following steps:

1. One minute rinse with 0.12% chlorhexidine in order to lower the microbial load of the oral cavity
2. Expose peri-apical x-rays with paralleling technique without removing the prosthesis in order to facilitate the alignment (Fig 2)
3. Observe patient oral hygiene maneuvers, use of toothbrush, super floss and inter proximal devices
4. Remove/unscrew the hybrid prosthesis
5. Position the prosthesis on a desk or flat plane with the intaglio surface facing up
6. Take a picture of the intaglio surface of the prosthesis
7. Take a clinical picture of the edentulous arch right after the removal of the prosthesis
8. Apply plaque disclosing agent on the edentulous ridge
9. Show the patient the areas stained by the plaque disclosing agent.
10. Show the patient on a monitor the picture of the intaglio surface of the prosthesis to point out areas where home hygiene can improve.
11. Hand to the patient a printout of the picture of the prosthesis with areas with plaque and calculus highlighted with arrows to better communicate ad reiterate the importance of proper hygiene (Fig 3)
12. Probe dental implants circumferentially using a UNC 15 periodontal probe. Record bleeding on probing (BoP), presence of plaque and probing pocket depth (PPD) at four sites per implant. Asses the tone and consistency of the peri implant soft tissues.
13. Decontaminate oral mucosa, gingiva, cheeks and tongue with the use of supragingival tip and erythritol powder. Set the machine at 50% power, 100% irrigation, keep the tip at 5mm distance form the soft tissues and move it with short back and forth movements at an inclination of 30-60°.
14. Decontaminate secondary implant components. Remove plaque disclosing agent, biofilm and staining with the use of supragingival tip and erythritol powder. Set the machine at 60-100% power, 100% irrigation, keep the tip at 3-5mm distance from the implant component and move it with short back and forth movements at an inclination of 60-90°.
15. Subgingival biofilm removal depends on PPD. Each site is treated specifically. If a site has PPD <5mm, decontaminate with the use of supragingival tip and erythritol powder. Set the machine at 60% power, 100% irrigation, keep the tip at 5mm distance from the peri implant sulcus and move it with short back and forth movements at an inclination of 30-60° and never at 90°. Use the tip 5 seconds per site at most.

    If a site has PPD >5mm PPD< 10mm, decontaminated with the use of subgingival tip (Perioflow®) and erythritol powder. Set the machine at 20-50% power, 70-100% irrigation (the % depends on peri implant tissue firmness), insert the tip in the peri implant sulcus and move it with short back and forth movements in an apical-coronal direction and is maintain it as parallel as possible to the long axis of the implant. Use the tip 5 consecutive seconds per site at most.
16. Remove, if present, remaining calculus with ultrasonic tip
17. Apply plaque disclosing agent again to double check complete biofilm removal
18. If needed remove remaining biofilm
19. Clean and polish the hybrid prosthesis
20. Reposition/Screw the prosthesis verifying absence of concavities and non-polished areas
21. Review and reinforce oral hygiene instructions
22. Schedule next maintenance visit according to patient's susceptibility

Peri-implants sulci will be probed using a UNC 15 periodontal probe at four sites, mesial, distal, lingual/palatal and buccal and clinical parameters such as plaque index (PlI), probing depth (PD), bleeding on probing (BOP) and peri-implant suppuration (PS) will be recorded immediately after removal of the prosthesis and at one month of follow-up.

Plaque index (PlI) will be evaluated through the use of a disclosing solution, applied with a cotton bud, at the same 4 sites for each implant. Peri-implant bleeding on probing (BOP) will also be evaluated at the same 4 sites for each implant. For both PlI and BOP, values from 0 to 4 will be recorded, depending on the number of implant surfaces presenting plaque/bleeding, respectively. Peri-implant tissue-suppuration (PS) will dichotomously be assessed (present/absent).

The collection of the microbiological sample will be carried out according to the following procedures: the implant will be isolated by suction and the use of cotton rolls, in order to avoid contamination of saliva. Four sterile endodontic paper points will be inserted into the peri-implant sulcus of each implant, placing them in the mesial, distal, lingual/palatal and buccal sites and removed after 30 seconds with tweezers by placing them in a sterile plastic tube which will be sealed immediately. The same procedure will be performed for each implant.

Once the operation is completed, the tubes of each patient (one for each implant and each containing 4 paper points) will be sent for microbiological analysis. The samples will be sent to the Microbiology Laboratory of the Department of Surgical Sciences of the University of Cagliari, in order to analyze the presence of bacteria of the peri-implant sulci. DNA from crevicular fluid samples will then be isolated by centrifugation and analyzed by PCR (polymerase chain reaction). This biomolecular technique is based on an enzymatic reaction, in which a heat-resistant DNA polymerase (Taq Polymerase) catalyzes the specific amplification of known DNA sequences. This procedure will be performed before the hygiene protocol, immediately after and at one month of follow-up.

Power analysis was employed to determine the sample size by using a .05 significance level and a power of 90% based on an effect size of 0.25. Sample size of 130 implants (approximately 25/30 patients carrying implant supported hybrid prostheses) is required to detect significant difference between the parameters measured at the different time points using repeated measures ANOVA. Descriptive statistics will be calculated, including means, standard deviations, medians, and confidence intervals. Microbiological outcomes measured at baseline, immediately post-maintenance and one month will be analyzed using the one-way repeated measures ANOVA test, while the statistical analysis of the PD, BOP, PlI and PS measurements at baseline and one month will be analyzed using McNemar's test. The level of significance is established at 5% (p = 0.05), and the analysis will be carried out using statistical software (SPSS version 26, IBM).

ELIGIBILITY:
Inclusion Criteria:

* Patients with implant-supported hybrid prosthesis

Exclusion Criteria:

* chronic bronchitis or asthma
* major systemic illnesses (i.e. diabetes mellitus, cancer, HIV, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy)
* Intake of antibiotics or other medication taken within the previous 28 days that may affect the outcome of the study
* Confirmed or suspected intolerance to erythritol or chlorhexidine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical parameters | immediately after removal of the prosthesis
  plaque index (PlI)
Clinical parameters | one month of follow-up.
  plaque index (PlI)
Clinical parameters | immediately after removal of the prosthesis
  probing depth (PD)
Clinical parameters | at one month of follow-up.
  probing depth (PD)
Clinical parameters | immediately after removal of the prosthesis
  bleeding on probing (BOP)
Clinical parameters | at one month of follow-up.
  bleeding on probing (BOP)
Clinical parameters | immediately after removal of the prosthesis
  peri-implant suppuration (PS)
Clinical parameters | at one month of follow-up.
  peri-implant suppuration (PS)
Microbiological parameters | immediately after removal of the prosthesis
  Four sterile endodontic paper points will be inserted into the peri-implant sulcus of each implant, placing them in the mesial, distal, lingual/palatal and buccal sites and removed after 30 seconds with tweezers by placing them in a sterile plastic tube which will be sealed immediately. The samples will be sent to the Microbiology Laboratory in order to analyze the presence of bacteria of the peri-implant sulci.
Microbiological parameters | at one month of follow-up.
  Four sterile endodontic paper points will be inserted into the peri-implant sulcus of each implant, placing them in the mesial, distal, lingual/palatal and buccal sites and removed after 30 seconds with tweezers by placing them in a sterile plastic tube which will be sealed immediately. The samples will be sent to the Microbiology Laboratory in order to analyze the presence of bacteria of the peri-implant sulci.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Duilio Casula, AOU Cagliari, Monserrato, CA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared in a publication after the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be submitted for publication right after the analysis of the outcomes

REFERENCES:
- [Background] Cobb CM, Daubert DM, Davis K, Deming J, Flemmig TF, Pattison A, Roulet JF, Stambaugh RV. Consensus Conference Findings on Supragingival and Subgingival Air Polishing. Compend Contin Educ Dent. 2017 Feb;38(2):e1-e4. PMID 28156118
- [Background] Taschieri S, Weinstein R, Del Fabbro M, Corbella S. Erythritol-Enriched Air-Polishing Powder for the Surgical Treatment of Peri-Implantitis. ScientificWorldJournal. 2015;2015:802310. doi: 10.1155/2015/802310. Epub 2015 May 6. PMID 26065025
- [Result] Riben-Grundstrom C, Norderyd O, Andre U, Renvert S. Treatment of peri-implant mucositis using a glycine powder air-polishing or ultrasonic device: a randomized clinical trial. J Clin Periodontol. 2015 May;42(5):462-9. doi: 10.1111/jcpe.12395. Epub 2015 Apr 30. PMID 25851433
- [Result] Cha JK, Paeng K, Jung UW, Choi SH, Sanz M, Sanz-Martin I. The effect of five mechanical instrumentation protocols on implant surface topography and roughness: A scanning electron microscope and confocal laser scanning microscope analysis. Clin Oral Implants Res. 2019 Jun;30(6):578-587. doi: 10.1111/clr.13446. Epub 2019 May 7. PMID 31022305